CLINICAL TRIAL: NCT06840860
Title: Monkeypox Biology, Outcome, Transmission and Epidemiology (MBOTE) Study: Epidemiological and Pathophysiological Insights Through a Cross-sectional Survey (EPIC)
Brief Title: Epidemiological and Pathophysiological Insights Through a Cross-sectional Survey (EPIC)
Acronym: MBOTE-EPIC
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Manitoba (Other); Catholic University of Bukavu, Democratic Republic of Congo (Unknown); University of Bern (Other); Alliance for International Medical Action (Other); Institut de Recherche pour le Developpement (Other Government); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 1835/24
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Monkeypox (Mpox)
Keywords: Monkeypox; Poxviridae Infections; Democratic Republic of Congo; Infections; Virus Diseases; DNA Virus Infections
MeSH Terms: conditions — Mpox, Monkeypox; Poxviridae Infections; Infections; Virus Diseases; DNA Virus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples With DNA — Venous blood: A maximum 10mL tube blood will be taken by venipuncture from adult participants and children aged 5 and over, while dried blood drops (DBS) will be used for children under 5 and babies.
  Skin Lesion swab: Skin swabs will be collected following the standard operating procedures of the national program, INRB and CDC recommendations; the base of the lesion is swabbed with a dry sterile flocked nylon swab. A single swab is used for sampling at least two separate lesions in two different locations on the body
  Oropharyngeal swab: Dry, flocked nylon swabs are used to swab the middle part of the throat, just beyond the tongue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to better understand how mpox is spreading in the DRC, how it affects different groups of people, and how well vaccines protect against it. The study is designed as a cross-sectional survey, meaning researchers will collect and analyze data from patients diagnosed with mpox at a single point in time. It will also use a case-control approach, comparing people who test positive for the virus to those who test negative, to identify risk factors and evaluate the effectiveness of the vaccine.

DETAILED DESCRIPTION:
This study aims to better understand how mpox is spreading in the DRC, how it affects different groups of people, and how well vaccines protect against it. The study is designed as a cross-sectional survey, meaning researchers will collect and analyze data from patients diagnosed with mpox at a single point in time. It will also use a case-control approach, comparing people who test positive for the virus to those who test negative, to identify risk factors and evaluate the effectiveness of the vaccine.

The study is being conducted by Institut National de Recherche Biomédicale (INRB) in collaboration with several international partners, including the Institute of Tropical Medicine (ITM) in Belgium, Johns Hopkins University, the University of Manitoba, Médecins Sans Frontières (MSF), and other leading research institutions. The study is funded by organizations such as the European & Developing Countries Clinical Trials Partnership (EDCTP3) and the Belgian Federal Government.

The study will be carried out in the DRC, focusing on provinces that have been hit hardest by mpox outbreaks, including North Kivu, South Kivu, Maniema, Kinshasa, and Equateur. Participants will be recruited from hospitals and health centers that provide mpox testing and care.

What Will Happen During the Study?

* People with suspected mpox who come to a hospital or health center for testing will be invited to participate.
* Participants will answer questions about their symptoms, medical history, and possible exposure to the virus, including vaccination status.
* Biological samples (blood, throat swabs, and skin lesion swabs) will be collected and analyzed for mpox and other infections such as measles or chickenpox.
* Hospitalized patients will have additional data recorded about their recovery.

Key Study Goals

* Describe how mpox affects people in different parts of the DRC, including symptoms, risk factors, and how the virus spreads.
* Compare differences between two types of the virus (clades Ia and Ib) to understand whether one is more severe than the other.
* Assess the effectiveness of the mpox vaccine by comparing vaccination rates between infected and uninfected individuals.
* Identify risk factors for severe disease, complications, and death in mpox patients.
* Investigate co-infections (e.g., with measles or chickenpox) that might worsen the disease.
* Support mpox treatment and prevention efforts by training healthcare workers and improving real-time data sharing through an online platform.

ELIGIBILITY:
Inclusion Criteria:

* Apply to be tested for VMPX at HGR or another test center.
* Patients of all ages and sexes. However, minors under the age of 12 are excluded from questions on sex life.
* The patient or his/her culturally acceptable representative is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will take place in the DRC, in the provinces most affected by mpox in recent months, namely North Kivu, South Kivu, Maniema, Kinshasa and Equateur. The study could be extended to other provinces, depending on the dynamics of the epidemic and research needs. Participants will be recruited from general referral hospitals (HGR) and from referral health centers (CSR) or health centers (CS) in the most affected areas, which provide mpox screening and management services.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical Manifestations of Mpox | 2 years
  The frequency and distribution of clinical symptoms and disease severity in confirmed mpox cases. (Percentage of cases presenting each symptom (e.g., fever, rash, lymphadenopathy)
Sociodemographic Characteristics of Confirmed Mpox Cases | 2 years
  The distribution of age, gender, occupation, and other demographic characteristics of confirmed mpox cases. (Mean/median values for continuous variables (e.g., age in years) and proportions for categorical variables (e.g., gender distribution, occupation)
Exposure Factors Among Mpox Cases | 2 years
  The percentage of cases reporting different exposure factors contributing to mpox transmission. ( Proportion of cases with specific exposure risks)
Modes of Transmission of Mpox | 2 years
  The relative contribution of different modes of transmission to the spread of mpox in the studied population. (Proportion of cases attributed to specific transmission routes)

SECONDARY OUTCOMES:
Proportion of Mpox Cases Among Individuals with and without Prior Orthopoxvirus Vaccination | 2 years
  This measure assesses the protective effect of prior vaccination against mpox by comparing vaccination coverage among PCR-confirmed cases versus unconfirmed suspected cases in a test-negative case-control study. The primary metric is the odds ratio (OR) of prior vaccination among cases versus controls, with vaccine efficacy (VE) calculated as VE = 1 - OR.
Regional Variability in Clinical Manifestations of Mpox | 2 years
  Comparison of the frequency and distribution of clinical symptoms and disease severity in confirmed mpox cases across different regions of the DRC.
Regional Variability in Sociodemographic Characteristics of Mpox Cases | 2 years
  Comparison of sociodemographic factors such as age, gender, occupation, and household composition among confirmed mpox cases in different regions.
Regional Variability in Exposure Factors for Mpox | 2 years
  Comparison of reported exposure factors (e.g., human contact, animal exposure) among mpox cases in different regions of the DRC.
Regional Variability in Modes of Mpox Transmission | 2 years
  Comparison of the distribution of transmission modes in different regions, identifying dominant transmission pathways.
Differences in Clinical Symptoms Between Mpox Clades Ia and Ib | 2 years
  The frequency of clinical symptoms will be compared between infections caused by Clade Ia and Clade Ib, based on genomic sequencing data.
Comparison of Disease Severity Between Mpox Clades Ia and Ib | 2 years
  The severity of mpox disease will be assessed and compared between Clade Ia and Clade Ib infections. Severity classification will follow standardized clinical definitions.
Comparison of Mpox Transmission Routes Between Clade Ia and Clade Ib Cases | 2 years
  Transmission modes will be compared between cases of Clade Ia and Clade Ib to identify potential differences in transmission dynamics.
Risk Factors for Severe Mpox Outcomes, Including Hospitalization and Mortality | 2 years
  This measure evaluates predictors of severe disease, including underlying comorbidities, demographic risk factors, and exposure history. It analyzes hospitalization rates, complications, and case fatality rates among mpox-positive patients.
Proportion of Mpox Cases with Co-infections Detected by PCR | 2 years
  This measure determines the prevalence of co-infections (e.g., measles, varicella, bacterial infections) among confirmed mpox cases, using PCR testing for other viral pathogens.
Estimating the Risk of Complications and Mortality in Mpox Cases | 2 years
  This measure quantifies the proportion of confirmed mpox cases that develop complications or result in fatality. A multivariate analysis will be conducted to identify independent predictors of severe disease progression.

CONTACTS AND LOCATIONS:
Locations (2):
- Democratic Republic of the Congo (2):
  - Masina Mpox Treatment Center, Kinshasa, Masina
  - Masina Mpox Treatment Center, Kinshasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brosius I, Vakaniaki EH, Mukari G, Munganga P, Tshomba JC, De Vos E, Bangwen E, Mujula Y, Tsoumanis A, Van Dijck C, Alengo A, Mutimbwa-Mambo L, Kumbana FM, Munga JB, Mambo DM, Zangilwa JW, Kitwanda SB, Houben S, Hoff NA, Makangara-Cigolo JC, Kinganda-Lusamaki E, Peeters M, Rimoin AW, Kindrachuk J, Low N, Katoto PDMC, Malembaka EB, Amuasi JH, Tshiani-Mbaya O, Kambaji DM, Kojan R, Kacita C, Mukadi-Bamuleka D, Ahuka-Mundeke S, Vercauteren K, Wawina-Bokalanga T, Muyembe-Tamfum JJ, Nundu SS, Liesenborghs L, Mbala-Kingebeni P. Epidemiological and clinical features of mpox during the clade Ib outbreak in South Kivu, Democratic Republic of the Congo: a prospective cohort study. Lancet. 2025 Feb 15;405(10478):547-559. doi: 10.1016/S0140-6736(25)00047-9. Epub 2025 Jan 29. PMID 39892407
- See also: MBOTE Consortium Website — https://www.mbote-mpox.com/